Cover page

May 1, 2016

NCT number NCT03171688

Official Title: Risk Factors for Nausea and Vomiting After Cesarean

Internal study ID: NVPOCesarianasGabriel2017





## INFORMED CONSENT

You are being invited to participate "Risk Factors for Nausea and Vomiting after Cesarean" study. You will receive all explanations you need before we start the research and we assure you that your name will not be shown and we will guarantee confidentiality by hiding any information which would identify you.

You will participate by answering some questions at Hospital Universitário de Brasília. The objective of this study is to find out what are the risk factors for nausea and vomiting after cesarean. You can refuse to participate this study with no personal disadvantage, we ensure that you may drop your consent anytime.

Your participation is voluntary, by that we mean that you will receive no money or advantage for the fact of participating the study.

The principal investigator will inform you of any unexpected or bad event you suffer due to participating. The results of this study will be published in our hospital's homepage, in a medical periodic as an article and may be cited by other articles or lectures about cesareans.

We plan to share all individual data with no identification variables (such as name or hospital register number) for transparency reasons, as a datasheet.

If you have any doubt related to this study, please ask doctor Gabriel Magalhaes Nunes Guimaraes from Hospital Universitario de Brasília, telephone number: 2028-5558, from 7am to 7pm, monday to friday.

This study was approved by the Ethics Comitee of Faculdade de Medicina da Universidade de Brasília. Any questions about this informed consent or your personal rights may be asked to them, telephone: 3107-1918 or by e-mail: cepfm@unb.br.

This Consent was print twice, one copy will be yours and the other will be hold by the investigator.

| Name / signature |
|------------------------|
| Principal investigator |
| Name / signature |